CLINICAL TRIAL: NCT06040541
Title: Phase 1/1b, Multicenter, Open-Label, Study of RMC 9805 in Participants With Advanced KRASG 12D-Mutant Solid Tumors
Brief Title: Study of RMC-9805 in Participants With KRAS G12D-Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-9805-001
Record Dates: First submitted 2023-08-31; First posted 2023-09-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Ductal Adenocarcinoma (PDAC); Advanced Solid Tumors
Keywords: KRAS G12D (ON); NSCLC; CRC; PDAC; Non-small Cell Lung Cancer; Lung Cancer; Colorectal Cancer; Colon Cancer; Pancreatic Cancer; Metastatic Cancer; Pancreatic Ductal Adenocarcinoma; Pancreatic Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; KRAS; Colonic Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Lung Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: The monotherapy arm of RMC-9805; the combination arm of RMC-9805 plus RMC-6236
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RMC-9805 monotherapy arm (Experimental): Dose exploration and dose expansion
  Interventions: Drug: RMC-9805
- RMC-9805 plus RMC-6236 combination arm (Experimental): Dose exploration and dose expansion
  Interventions: Drug: RMC-9805; Drug: RMC-6236

INTERVENTIONS:
Drug: RMC-9805 — Oral Tablets
Drug: RMC-6236 — Oral Tablets
  Arms: RMC-9805 plus RMC-6236 combination arm

SUMMARY:
This study is to evaluate the safety and tolerability of RMC-9805 as monotherapy and in combination with RMC-6236 in adults with KRAS G12D-mutant solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/1b study of RMC-9805, a selective and orally bioavailable KRAS G12D(ON) inhibitor, in subjects with KRASG12D-mutant solid tumors to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary clinical activity. The study consists of two arms: RMC-9805 monotherapy arm and RMC-9805 plus RMC-6236 combination arm. Both arms consist of two parts: Part 1- dose exploration and Part 2- dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented, locally advanced or metastatic solid tumor with a KRAS G12D-mutation
* Received and progressed or been intolerant to prior standard therapy (including targeted therapy) appropriate for tumor type and stage
* ECOG performance status 0 or 1
* Adequate organ function

Exclusion Criteria:

* Primary central nervous system (CNS) tumors
* Known or suspected leptomeningeal or active brain metastases or spinal cord compression
* Known or suspected impairment of gastrointestinal function that may prohibit ability to swallow or absorb an oral medication
* Participant was previously treated with an investigational KRAS G12D inhibitor, pan- or multi-RAS inhibitor, or had prior therapy with any direct RAS-targeted therapy (eg, degraders and inhibitors)

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 3 years
  Incidence and severity of treatment-emergent Adverse Events (AEs) and serious AEs and clinically significant changes in laboratory values, ECGs, and vital signs
Dose Limiting Toxicities | 21 days
  Number of participants with Dose Limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
Maximum Observed Blood Concentration (Cmax) of RMC-9805 as monotherapy and in combination with RMC-6236, and Cmax of RMC-6236 in combination with RMC-9805 | up to 21 weeks
  Cmax
Time to Reach Maximum Blood Concentration (Tmax) of RMC-9805 as monotherapy and in combination with RMC-6236, and Tmax of RMC-6236 in combination with RMC-9805 | up to 21 weeks
  Tmax
Area Under Blood Concentration Time Curve (AUC) of RMC-9805 as monotherapy and in combination with RMC-6236, and AUC of RMC-6236 in combination with RMC-9805 | up to 21 weeks
  AUC
Ratio of accumulation of RMC-9805 from a single dose to steady state with repeated dosing as monotherapy and in combination with RMC-6236, and ratio of accumulation of RMC-6236 in combination with RMC-9805 | up to 21 weeks
  accumulation ratio
Elimination Half-Life (t1/2) of RMC-9805 as monotherapy and in combination with RMC-6236, and t1/2 of RMC-6236 in combination with RMC-9805 | up to 21 weeks
  t1/2
Overall Response Rate (ORR) | up to 3 years
  Assess per RECIST v1.1
Duration of Response (DOR) | up to 3 years
  Assess per RECIST v1.1
Disease Control Rate (DCR) | up to 3 years
  Assess per RECIST v1.1
Time to Response (TTR) | up to 3 years
  Assess per RECIST v1.1
Progression-Free Survival (PFS) | up to 3 years
  Assess per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (17):
- United States (17):
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Hospital (Yale University), New Haven, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - Lee Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - START, San Antonio, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia

REFERENCES:
- [Derived] Weller C, Burnett GL, Jiang L, Chakraborty S, Zhang D, Vita NA, Dilly J, Kim E, Maldonato B, Seamon K, Eilerts DF, Milin A, Marquez A, Spradlin J, Helland C, Gould A, Ziv TB, Dinh P, Steele SL, Wang Z, Mu Y, Chugh S, Feng H, Hennessey C, Wang J, Roth J, Rees M, Ronan M, Wolpin BM, Hahn WC, Holderfield M, Wang Z, Koltun ES, Singh M, Gill AL, Smith JAM, Aguirre AJ, Jiang J, Knox JE, Wildes D. A neomorphic protein interface catalyzes covalent inhibition of RASG12D aspartic acid in tumors. Science. 2025 Jul 24;389(6758):eads0239. doi: 10.1126/science.ads0239. Epub 2025 Jul 24. PMID 40705880
- [Derived] Cregg J, Edwards AV, Chang S, Lee BJ, Knox JE, Tomlinson ACA, Marquez A, Liu Y, Freilich R, Aay N, Wang Y, Jiang L, Jiang J, Wang Z, Flagella M, Wildes D, Smith JAM, Singh M, Wang Z, Gill AL, Koltun ES. Discovery of Daraxonrasib (RMC-6236), a Potent and Orally Bioavailable RAS(ON) Multi-selective, Noncovalent Tri-complex Inhibitor for the Treatment of Patients with Multiple RAS-Addicted Cancers. J Med Chem. 2025 Mar 27;68(6):6064-6083. doi: 10.1021/acs.jmedchem.4c02314. Epub 2025 Mar 8. PMID 40056080